CLINICAL TRIAL: NCT00146653
Title: A Comparison of Heparin Management Strategies in Children Undergoing Cardiopulmonary Bypass.
Brief Title: Heparin Management During Cardiopulmonary Bypass in Children
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nina Guzzetta, M.D., Assistant Professor of Anesthesiology, Emory University
Other Study IDs: 286-2005
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Primary Condition: Heart Defects Requiring Surgery With CPB
Keywords: pediatrics; cardiopulmonary bypass; surgery

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is being collected to obtain Xa results.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xa: An additional 20 patients will be enrolled to address the validation of heparin concentrations calculated by the Hepcon machine with laboratory-measured heparin concentrations. These patients will not be randomized and therefore will not receive an intervention. .

SUMMARY:
We propose a comparison between between our standard ACT based heparin management protocol for children undergoing CPB and a patient-specific heparin concentration-based heparin management protocol. We hypothesize that a heparin concentration-based anticoagulation management protocol during CPB in children will result in more effective attenuation of hemostatic activation as reflected by decreased levels of thrombin formation and, ultimately, better preservation of hemostasis postoperatively.

An additional 20 patients will be enrolled to address the validation of heparin concentrations calculated by the Hepcon machine with laboratory-measured heparin concentrations. These patients will not be randomized and therefore will not receive an intervention.

DETAILED DESCRIPTION:
40 patients will be randomly assigned to either the traditional heparin management group or the intervention group. The traditional group will be treated with an initial heparin dose of 400 units/kg and the standard amount of heparin, as dictated by the circuit size, will be added to the CPB circuit prime. An ACT target value of 480 seconds will be maintained throughout the bypass period. Should the ACT fall below 480 seconds,additional boluses of 100 units/kg of heparin will be given until the ACT returns to the target value. At the end of CPB, heparin will be neutralized by the standard reversal of 4 mg/kg of protamine.

An additional 20 patients will be enrolled to address the validation of heparin concentrations calculated by the Hepcon machine with laboratory-measured heparin concentrations. These patients will not be randomized and therefore will not receive an intervention.

For the intervention group, a heparin dose (HDR) response assay will be performed prior to surgical incision by the Hepcon instrument. The hepcon machine performs a patient-specific HDR assay based on body surface area, and determines a projected heparin concentration required by that patient to achieve an ACT of 480 seconds. The HDR assay provides the initial dose of heparin to give the patient as well as the amount of heparin to be added to the CPB circuit. Additional heparin doses as determined by the hepcon instrument will be administered as needed if the patient's heparin concentration falls below the projected reference concentration. The hepcon instrument will also calculate the protamine dose needed to reverse heparin at the end of CPB.

For comparison between groups, an assay using the hepcon machine to measure whole blood heparin concentration and an ACT will be obtained for each patient at the following intervals: after the initial heparin dose, 30 minutes after the initiation of CPB, the start of rewarming and immediately prior to the discontinuation of CPB. A sample for anti-factor Xa activity will also be obtained at each of the above time intervals to validate the heparin concentration determined by the hepcon machine to a laboratory measured value. Blood samples for biochemical markers of hemostatic activation will be collected from all patients before the initiation of CPB after the administration of the initial heparin dose and after the conclusion of CPB before protamine infusion. The following biochemical markers of hemostatic activation will be measured: prothrombin fragment 1.2, fibrinopeptide A, free tissue factor pathway inhibitor, factor V, factor VIII, and beta-thromboglobulin. The following measures of clinical outcome will also be recorded: amount of blood products transfused after protamine administration, time between the administration of protamine to leaving the operating room, 24-hour chest tube drainage, first post-operative weight, time to extubation and duration of ICU stay.

Additional 20 patients: These additional 20 patients will be enrolled to provide further validation of the Hepcon-measured heparin concentrations with the laboratory-measured heparin concentrations (anti-factor Xa activity). A blood sample will be obtained for a heparin dose response (HDR) assay prior to surgical incision Samples will also be obtained to measure a heparin concentration by the Hepcon machine and by anti-factor Xa activity at two time periods: after the initial heparin dose and immediately prior to discontinuation of CPB. In addition, these 20 patients will also have an ACT test analyzed by the Hepcon machine after protamine is given.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective cardiac surgical procedures requiring CPB at Children's Healthcare of Atlanta at Egleston.
2. Patients less than 6 months old.
3. Parent/legal guardian willing to sign consent. -

Exclusion Criteria:

1. Patients presenting for emergency surgery.
2. Patients treated preoperatively with anticoagulant therapy.
3. Patients treated with antifibrinolytics during their cardiac surgery.
4. Parent/legal guardian unwilling or unable to sign consent. -

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be obtained from the patient's of Children's Healthcare of Atlanta at Egleston. These patients will be obtained from the pre-operative clinc, the Cardiac Intensive Care Unit or the Cardiac Stepdown unit.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Xa sample is being collected to validate the results from the Hepcon Assay. The Hepcon results are being compared to the Hemochron and iStat ACT results. | The Xa sample is being collected before the initiation of cardiopulmonary bypass and immediately prior to the discontinuation of cardiopulmonary bypass.

SECONDARY OUTCOMES:
Transfusion requirements and patient bleeding postoperatively. | Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Guzzetta, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Culliford AT, Gitel SN, Starr N, Thomas ST, Baumann FG, Wessler S, Spencer FC. Lack of correlation between activated clotting time and plasma heparin during cardiopulmonary bypass. Ann Surg. 1981 Jan;193(1):105-11. doi: 10.1097/00000658-198101000-00017. PMID 6970015
- [Background] Horkay F, Martin P, Rajah SM, Walker DR. Response to heparinization in adults and children undergoing cardiac operations. Ann Thorac Surg. 1992 May;53(5):822-6. doi: 10.1016/0003-4975(92)91444-e. PMID 1570978